CLINICAL TRIAL: NCT05059288
Title: Usability and Performance of a Non-invasive Ventilation Mask. A Prospective Cohort.
Brief Title: NIV Mask Assessment of Usability and Performance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CIA 291
Record Dates: First submitted 2021-09-06; First posted 2021-09-28 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Investigation Mask (Experimental): Non invasive ventilation mask
  Interventions: Device: Investigational Non Invasive Ventilation Mask

INTERVENTIONS:
Device: Investigational Non Invasive Ventilation Mask — Oronasal non invasive ventilation mask

SUMMARY:
Assessment of usability, perceived comfort and performance of a NIV mask in the hospital environment.

DETAILED DESCRIPTION:
50 participants admitted for NIV therapy will have the investigation mask fitted. The doctors and nurses assigned to the participants care will complete a subjective evaluation on how the mask performs compared to the standard of care mask. Some therapy settings and demographics will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Admitted and indicated for non invasive ventilation therapy
* Assessed for capacity to consent and consent process documented
* Fits the investigation mask
* Aged 18 year or older

Exclusion Criteria:

- Contraindicated for non invasive ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-10-28 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Perceived mask performance | During the intervention
  Three point visual analogue scale on preference 1 = Worse, 2 = Same, 3 = Better

CONTACTS AND LOCATIONS:
Overall Officials: Robert Martynoga, Principal Investigator — Waikato Hospital

IPD SHARING:
Plan to Share IPD: No